CLINICAL TRIAL: NCT06286059
Title: Protective Efficacy of Phentolamine in Patients at High Risk of Contrast-Associated Acute Kidney Injury After Complex Percutaneous Coronary Intervention
Brief Title: Efficacy of Phentolamine in Prevention of Contrast-Associated Acute Kidney Injury After Complex PCI
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohammed Soliman Mostafa Mohammed, Doctor, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Phentolamine for CA-AKI
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: CA-AKI - Contrast-Associated Acute Kidney Injury; Coronary Artery Disease; Acute Coronary Syndrome; Adrenergic Receptor Antagonist Adverse Reaction
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Phentolamine

STUDY DESIGN:
Intervention Model Description: Randomised controlled clinical trial
Who Masked: Participant
Masking Description: Single Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients will receive conventional management including high dose atorvastatin and isotonic (0.9%) saline intravenous (IV) infusion at a rate of 1 ml/kg/hr for 12 hours or reduced to 0.5 ml/kg/hr if the patient's LVEF < 40% or overt heart failure.
- Phentolamine group (Experimental): In addition to the conventional management, patients will receive phentolamine infusion.
  Interventions: Drug: Phentolamine

INTERVENTIONS:
Drug: Phentolamine — In addition to the conventional management, patients will receive phentolamine (Rogitamine; Egypharma) infusion at a rate of 0.5 μgm/kg/min for the first 15 minutes after a bolus dose of 5 mg. If significant hemodynamic change occurred, the infusion then will be discontinued and the patient will be excluded. Otherwise, the dose will be uptitrated gradually 0.5-2 ugm/kg/min and the infusion will be continue for 12 hours.
  Other Names: Rogitamine
  Arms: Phentolamine group

SUMMARY:
To evaluate the efficacy and safety of phentolamine in prevention of CA-AKI following complex PCI in patients at high risk of CA-AKI.

DETAILED DESCRIPTION:
Coronary angiography is accepted as the gold standard diagnostic procedure in the management of coronary artery disease (CAD). It involves the visualization of the coronary arteries using contrast dye and dynamic X-ray imaging and allows for the identification of suitable lesions for percutaneous coronary intervention (PCI). PCI has more importance when performed as an emergency procedure during acute coronary syndromes (ACS) providing immediate relief of symptoms, preventing myocardial damage and reducing mortality rates despite its potential complications. These complications varies in its incidence including arrhythmias, coronary dissection, bleeding at the access site, allergy to contrast agent and kidney injury with varying risk on patient condition.

Contrast-associate acute kidney injury (CA-AKI), formerly termed contrast-induced nephropathy (CIN), is a significant complication of PCI and the third most common cause of renal failure in hospitalized patients. It is defined as a rise in creatinine of ≥ 50% of baseline or 0.3 mg/dL from the pre-contrast value within 48-72 hours of intravascular administration of a contrast medium, which is usually reversible acute kidney injury. The development of CA-AKI despite successful percutaneous coronary procedures is associated with prolonged hospitalization, an increase in health expenditure, and increased short and long-term mortality for most patients. Therefore, early risk prediction and management is crucial.

Over the past few decades, a number of risk scores have been introduced to predict contrast-associated acute kidney injury after PCI. The most commonly used is Mehran score that was introduced in 2004 for its simplicity and availability but it excluded patients with acute myocardial infarction. However, it recently updated with larger population and more emphasis on patient's ACS presentation and procedural features and reintroduced in 2021 as Mehran 2 CA-AKI Risk Score.

Exact pathophysiological mechanism of CA-AKI is not known and includes complex cascades of events. The most important elements of pathophysiological mechanism of CA-AKI seem to be the medullary hypoxia due to contrast-induced medullary vasoconstriction and direct renal tubular cytotoxicity, in addition to oxidative stress and the increase in blood and renal tubular viscosity which are complementary events that further exacerbates CA-AKI.

Several clinical interventions aimed to reduce the incidence of CA-AKI targeting various aspects of the pathophysiology including volume expansion with intravenous fluid, administration of N-acetylcysteine, sodium bicarbonate, vitamin E, statins and vasodilator agents with different protective efficacy but only few of them had been approved for clinical practice.

Vasodilators agents like nicorandil showed a statistically significant lower odds of developing CA-AKI with periprocedural hydration and the vasodilator agent nicorandil versus periprocedural hydration only (OR: 0.173). Also, a recent clinical trial has demonstrated encouraging results regarding the renoprotective effects of phentolamine in chronic coronary syndrome following PCI with odds ratio 0.04 of CA-AKI in phentolamine group in comparison to control group.

Phentolamine, a non-selective alpha-adrenergic antagonist, is primarily used for the treatment of conditions involving excessive sympathetic activity. While it is not a commonly used medication in the management of CAD, it used in various cardiovascular urgent conditions as in hypertensive crisis and in the treatment of cocaine-induced ACS which counteract the excessive sympathetic stimulation and reduce peripheral vascular resistance in conjunction with other treatments to alleviate symptoms and improve hemodynamics with less incidence of tachycardia associated with other vasodilators e.g. nitroglycerin.

This clinical trial will investigate the potential of phentolamine as a renoprotective agent following complex PCI by evaluating the impact of phentolamine on renal outcomes and its safety which may significantly impact clinical practice by guiding the use of phentolamine as an adjuvant therapy, ultimately improving patient outcomes and reducing the burden of CA-AKI in high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to CCU with CAD.
* Patients underwent successful complex PCI defined as multivessel disease, more than two lesions, high coronary lesion complexity, chronic total occlusion, lesion length >30 mm, or bifurcation.
* Patients at high or very high risk for CA-AKI based on Mehran-2 CA-AKI Risk Score (Model 2).

Exclusion Criteria:

* Patients with end stage renal disease on regular dialysis.
* Patients with failed PCI revascularization.
* Patients presented with STEMI and underwent primary PCI.
* Patients presented with high risk NSTEMI defined as elevated cardiac enzymes with chest pain refractory to medications and/or dynamic ST changes.
* Patients presented with cardiogenic shock.
* Patients presented with any degree of heart block.
* Patients with of history of asthma or hypersensitive for phentolamine.
* Patients on α-blockers, barbiturates or antipsychotic treatment.
* Patients intolerant to phentolamin with significant hemodynamic changes defined as >20% drop of systolic blood pressure (SBP) or >20% increase of heart rate (HR) after loading dose of phentolamine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of CA-AKI | 3 days post-PCI
  A rise in creatinine of ≥ 50% of baseline or 0.3 mg/dL from the pre-contrast value within 48-72 hours of intravascular administration of a contrast medium.

SECONDARY OUTCOMES:
Peak of serum creatinine elevation | 7 days
  Maximum level of serum creatinine reached in patients who developed CA-AKI
Duration of CA-AKI | 14 days
  Duration of CA-AKI in patients who developed CA-AKI
Change in HR | 12 hours post-PCI
  Change in heart rate
Change in SBP | 12 hours post-PCI
  Change in systolic blood pressure
Change in DBP | 12 hours post-PCI
  Change in diastolic blood pressure
Urine output | 12 hours post-PCI
  Urine output per hour post-PCI
Rate of RRT | 7 days
  Rate of patients needed renal replacement therapy
Rate of MACE | 30 days post-PCI
  Composite rate of myocardial injury, non-fatal MI, non-fatal stroke, and all-cause mortality.
Rate of rehospitalization | 30 days post-PCI
  Unplanned hospitalization during the first month post-PCI
Duration of hospitalization | 14 days
  Duration of hospitalization post-PCI until hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Sadek, Professor, Study Chair — Helwan University; Arafa Gomaa, MD, Study Director — Helwan University
Locations (1):
- Badr university hospital, Badr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Master sheet of decoded data of the participants
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months after end of the study duration
Access Criteria: Supporting information will be added to the original study during publishing

REFERENCES:
- [Background] Hamila MA, El Ghawaby H, Zaki M, Soliman M, Gabr K. Association of periprocedural phentolamine infusion with favorable outcome in patients with chronic kidney disease and chronic coronary syndrome undergoing coronary catheterization: a prospective randomized controlled pilot study. BMC Nephrol. 2022 Dec 31;23(1):416. doi: 10.1186/s12882-022-03050-9. PMID 36585656
- [Background] Kelesoglu S, Yilmaz Y, Elcik D, Cetinkaya Z, Inanc MT, Dogan A, Oguzhan A, Kalay N. Systemic Immune Inflammation Index: A Novel Predictor of Contrast-Induced Nephropathy in Patients With Non-ST Segment Elevation Myocardial Infarction. Angiology. 2021 Oct;72(9):889-895. doi: 10.1177/00033197211007738. Epub 2021 Apr 8. PMID 33827291
- [Background] Lu Y, Wang Y, Zhou B. Predicting long-term prognosis after percutaneous coronary intervention in patients with acute coronary syndromes: a prospective nested case-control analysis for county-level health services. Front Cardiovasc Med. 2023 Dec 4;10:1297527. doi: 10.3389/fcvm.2023.1297527. eCollection 2023. PMID 38111892
- [Background] Mehran R, Owen R, Chiarito M, Baber U, Sartori S, Cao D, Nicolas J, Pivato CA, Nardin M, Krishnan P, Kini A, Sharma S, Pocock S, Dangas G. A contemporary simple risk score for prediction of contrast-associated acute kidney injury after percutaneous coronary intervention: derivation and validation from an observational registry. Lancet. 2021 Nov 27;398(10315):1974-1983. doi: 10.1016/S0140-6736(21)02326-6. Epub 2021 Nov 15. PMID 34793743
- [Background] Ozkok S, Ozkok A. Contrast-induced acute kidney injury: A review of practical points. World J Nephrol. 2017 May 6;6(3):86-99. doi: 10.5527/wjn.v6.i3.86. PMID 28540198
- [Background] Walker H, Guthrie GD, Lambourg E, Traill P, Zealley I, Plumb A, Bell S. Systematic review and meta-analysis of prophylaxis use with intravenous contrast exposure to prevent contrast-induced nephropathy. Eur J Radiol. 2022 Aug;153:110368. doi: 10.1016/j.ejrad.2022.110368. Epub 2022 May 23. PMID 35636024